CLINICAL TRIAL: NCT01850056
Title: Prospective, Multi-center and Randomized Controlled Clinical Study to Verify Effectiveness and Safety of Drug-eluting Balloon in PTA Procedure (AcoArt I Study)
Brief Title: AcoArt Ⅰ / SFA China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: acotec-02
Record Dates: First submitted 2013-04-27; First posted 2013-05-09 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2015-12

CONDITIONS: Peripheral Artery Disease
Keywords: drug eluting balloon catheter
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- drug eluting balloon catheter (Experimental): use drug eluting balloon catheter to inflate the stenosis or occlusion in superficial femoral artery(SFA) and/or popliteal artery
  Interventions: Device: drug eluting balloon catheter (trade name: Orchid)
- common balloon catheter(uncoated drug) (Active Comparator): use common balloon catheter to inflate stenosis or occlusion in SFA and/or popliteal artery
  Interventions: Device: common percutaneous transluminal angioplasty balloon catheter (trade name: Admiral)

INTERVENTIONS:
Device: drug eluting balloon catheter (trade name: Orchid)
  Other Names: drug eluting dilation catheter
  Arms: drug eluting balloon catheter
Device: common percutaneous transluminal angioplasty balloon catheter (trade name: Admiral)
  Other Names: common PTA catheter
  Arms: common balloon catheter(uncoated drug)

SUMMARY:
The purpose of this study is to determine whether DEB is more effective than common PTA balloon in long-term vessel patency and inhibiting restenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Patients with peripheral artery disease (PAD), with Rutherford classification between 2 and 5
* an occlusion or a minimum grade of stenosisPrimary over 70% in the superficial femoral artery an /or the popliteal artery
* Total length of treat lesion(s)is less or equal to 40cm
* signed Patient informed consent form

Exclusion Criteria:

* plasma Cr level greater than 150 umol/L in patients
* patients with acute thrombosis requiring lysis or thrombectomy
* patient with a lysis or an lower limb intervention as a therapy within the last 6 weeks
* patient requiring intervention in both lower limbs at the same time
* target lesion can't be cross by the guide wire
* distal outflow through less than one lower leg vessel
* known hypersensitivity to aspirin, heparin, clopidogrel,paclitaxel, contrast medium, etc.
* patients participating in another clinical trials with interfere with this trial in the past 3 months
* pregnancy and lactating woman
* untreatable bleeding diatheses
* other diseases, such as cancer, liver disease, or cardiac insufficiency, which may lead to protocol violations or markedly shorten a patients's life expectancy(less than 2 years)
* patients unable or unwilling to participate this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Late Lumen Loss | 6 months
  measure difference of the MLD(minimal lumen diameter) at 0 time and 6 months

SECONDARY OUTCOMES:
Minimal lumen diameter (MLD) | 6 months
  measure minimal lumen diameter (MLD) of target lesion
Restenosis rate of target vessel | 6 months, 12 months, 18 months, 24months
  stenosis over 50% is defined as restenosis
target lesion revascularization | 6 months, 12 months, 18 months, 24 months
  target lesion revascularization is defined as any reintervention of artery bypass graft surgery involving the target lesion
change in Rutherford stage | 6 months, 12 months, 18 months, 24 months
  based the following definition of Rutherford stage, evaluate the stage of patient. Then compare the stage of patient just after procedure and 6 months after treatment
  Stage clinical symptom
  0 asymptomatic
  1. mild claudication
  2. moderate claudication
  3. severe claudication
  4. ischemic rest pain
  5. minor tissue loss
  6. ulceration or gangrene
change in ankle brachial index(ABI) | 6 months
  change in ankle brachial index(ABI) compared to pretreatment
major amputation | 6 months, 12 months, 18 months, 24 months
  major amputation at the index limb(major amputation is defined as an amputation above the foot)
Death | 12 months, 18 months, 24 months
  death of any cause

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Xiyuan Hospital CACMS, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The second Hospital Of Hebei University, Shijiazhuang, Hebei
  - The First Affiliated Hospital, Dalian Medical University, Dalian, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital ShangHai Jiaotong University School Of Medicine, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Ren H, Liu J, Zhang J, Zhuang B, Fu W, Wu D, Wang F, Zhao Y, Guo P, Bi W, Wang S, Guo W. Five-Year Outcomes of Post-Drug-Coated Balloon Angioplasty Dissection in Complex Femoropopliteal Artery Disease. Int J Gen Med. 2021 Aug 5;14:4197-4207. doi: 10.2147/IJGM.S316916. eCollection 2021. PMID 34385840
- [Derived] Sun G, Liu J, Jia S, Zhang J, Zhuang B, Jia X, Fu W, Wu D, Wang F, Zhao Y, Guo P, Bi W, Wang S, Guo W; AcoArt I Trial Investigators. Comparison of drug-coated balloon angioplasty versus uncoated balloon angioplasty in treatment of total occlusions with severe femoropopliteal lesions: An additional analysis from the AcoArt I study. Vascular. 2021 Jun;29(3):340-349. doi: 10.1177/1708538120953663. Epub 2020 Sep 9. PMID 32903168